CLINICAL TRIAL: NCT00193960
Title: A Comparison Between Superior and Inferior Ahmed Glaucoma Valve Implantation: Surgical Success and Complications
Brief Title: The Results of Ahmed Valve Operations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: In process
Record Dates: First submitted 2005-09-09; First posted 2005-09-19 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-09

CONDITIONS: Glaucoma
Keywords: Seton surgery, glaucoma, Ahmed valve, intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: 1) Intraocular pressure 2) visual acuity

SUMMARY:
Glaucoma drainage devices are usually placed in the superior quadrants. The superotemporal quadrant is usually the site of choice. However, when the upper fornix is scarred and especially when conjunctiva is two fibrotic to enable adequate coverage of tube with a scleral or other patch graft, some surgeons place the tube in one of inferior quadrants.

DETAILED DESCRIPTION:
Glaucoma drainage devices are usually placed in the superior quadrants. The superotemporal quadrant is usually the site of choice. However, when the upper fornix is scarred and especially when conjunctiva is two fibrotic to enable adequate coverage of tube with a scleral or other patch graft, some surgeons place the tube in one of inferior quadrants.

In the present study we will compare the outcome and complicatons of both the superior and the inferior approach for inserting Ahmed Valve implants.

ELIGIBILITY:
Inclusion criteria:

1. Patients at the ages of 20-85 on the date of the surgery
2. The indication for the surgery was: uncontrolled glaucoma with maximally tolerated medical therapy who did not or were not expected to respond to other surgical procedures than seton surgery.
3. Visual acuity of, at least, 20/800 before the operation.
4. Regular post operative follow ups, for at least 1 year.
5. Patients after corneal transplantation for whom the indication of valve implantation was uncontrolled glaucoma.

Exclusion Criteria:

1. A previous seton surgery in the operated eye
2. Uveitic glaucoma patients or history of uveitis in the operated or in the fellow eye.
3. Any inflammatory or ocular surface disease that could affect the healing of the conjunctiva after the surgery ( e.g: OCP)
4. Strabismus or complains of diplopia prior to the seton surgery.
5. Past history of retinal detachment surgery with scleral buckle in the operated eye
6. Past history of endophthalmitis in the operated eye.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1997-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Trope E Graham, MB, FRCSC, Study Director — University of Toronto, Department of Ophthalmology; Rony Rachmiel, M.D, Study Director — University of Toronto, Department of Ophthalmology
Locations (1):
- Department of Ophthalmology and visual sciences, Toronto Western Hospital,, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rachmiel R, Trope GE, Buys YM, Flanagan JG, Chipman ML. Ahmed glaucoma valve implantation in uveitic glaucoma versus open-angle glaucoma patients. Can J Ophthalmol. 2008 Aug;43(4):462-7. doi: 10.3129/i08-082. PMID 18711462